CLINICAL TRIAL: NCT07079332
Title: Structural Validity and Inter-rater Reliabitiliy of the Ataxia Trunk, Lower And Upper Extremity Scale (ATLAS)
Acronym: ATLASReVa
Status: Not yet recruiting | Type: Observational
Sponsor: Haute Ecole de Santé Vaud (Other)
Responsible Party: Principal Investigator, HESAV Health Research Unit, Lecturer, Haute Ecole de Santé Vaud
Other Study IDs: ATLAS_01; 16-M25 (Other Grant/Funding Number: Health Domain Scientific Committee of HES-SO University of Applied Sciences and Arts Western Switzerland); 2025-01498 (Other: Swissethics)
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Ataxia, Cerebellar; Ataxia, Gait; Ataxia, Motor; Ataxia; Ataxia, Spinocerebellar; Ataxias, Hereditary; Ataxia - Other
Keywords: Ataxia; Scale; Validity Study; reliability study; new scale
MeSH Terms: conditions — Cerebellar Ataxia; Gait Ataxia; Ataxia; Spinocerebellar Ataxias; Spinocerebellar Degenerations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ataxia patient: Presenting motor symtpoms of ataxia
  Interventions: Other: New Scale to evaluate ataxia motor symptoms

INTERVENTIONS:
Other: New Scale to evaluate ataxia motor symptoms — The Ataxia Trunk, Lower And upper extremity Scale (ATLAS) is a new scale. It differs from other Ataxia Scale by focusing on the assessment of coordination abilities of specific body segments: the trunk, lower limbs, and upper limbs.

SUMMARY:
Ataxia is a neurological disorder affecting coordination, caused by damage to the cerebellum, brainstem, or related pathways. It can be hereditary (e.g., Friedreich's ataxia) or acquired (e.g., multiple sclerosis, stroke). Though rare, ataxia significantly impacts quality of life and independence. Treatments are limited and mainly focus on multidisciplinary rehabilitation. Accurate assessment is essential, yet current tools like Scale for the Assessment and Rating of Ataxia (SARA) have limitations. This study aims to validate a new scale, named the Ataxia Trunk, Lower And upper extremity Scale (ATLAS), through Rasch analysis, to develop a shorter, reliable version. It will assess internal consistency, construct validity, and inter-rater reliability.

For the valitdity part, statistics will be used (1) to see if the different items of the scale are indeed different and complementary to each other, and (2) to compare the results of this scale with other scales already known and valid (SARA, Trunk Impairment Scale (TIS) and Functional Impairment Measurement(FIM)). Secondly, the investigators would like to know whether ATLAS is reliable. In this particular case, the reliability being assessed is inter-rater reliability, i.e. whether all raters give the same score on the items performed by the patient. To carry out such a study, 64 people will be needed to achieve these goals. Each person will complete the 20 items of the ATLAS scale, those of a trunk motor capacity assessment (TIS), and will evaluate his or her functional independence (FIM).

DETAILED DESCRIPTION:
Ataxia, derived from the Greek word ataxia meaning "disorder," is a neurological condition characterized by impaired coordination of oculomotor movements, upper limbs (UL), lower limbs (LL), and trunk, as well as dysarthria. Most of these symptoms lead to disturbances in postural control and gait. Ataxia may result from damage to the cerebellum, brainstem, and/or ascending pathways.

In addition to these motor impairments, vestibulocerebellar syndrome and cerebellar cognitive affective syndrome (also known as Schmahmann's syndrome) contribute to difficulties in regulating cognitive, motivational, and emotional states in affected individuals.

Ataxias are broadly classified into two main categories:

I) Hereditary or genetic ataxias, with an overall prevalence of approximately 2.7-38.35 per 100,000, include Friedreich's ataxia (autosomal recessive), other autosomal recessive ataxias (average prevalence of 3.3 per 100,000), and spinocerebellar ataxias (mostly autosomal dominant, average prevalence of 2.7 per 100,000).

II) Acquired ataxias, which may result from multiple sclerosis (MS; 100 per 100,000, with 10-50% showing signs of ataxia), stroke, traumatic brain injury (TBI), tumors, infections, vitamin deficiencies, or exposure to toxic substances such as alcohol, heavy metals, or medications.

Genetic ataxias affect men and women equally 1, whereas acquired ataxias show gender disparities depending on the underlying condition: MS affects approximately 1 male for every 4 females; stroke affects 1 male for every 1.28 females; TBI affects 3 males for every 1 female.

Across all types, ataxia affects approximately 1 in 10,000 individuals, making it a relatively rare condition. However, its impact on quality of life and employability is substantial, as it compromises mobility, independence, and the ability to perform daily activities. It increases reliance on healthcare professionals and reduces the quality of life of caregivers due to the growing burden. Ultimately, it also raises mortality risk. The average annual cost per patient was estimated at €18,776 in 2014. These psycho-socio-economic consequences justify scientific interest, particularly regarding treatment efficacy and appropriate assessment.

Treatments

Effective curative treatments are rare or nonexistent for most genetic ataxias. Only a few drugs, such as Riluzole and 4-Aminopyridine, may slightly slow disease progression or symptom expression. A Riluzole precursor, Triluzole, is currently undergoing phase III clinical trials. Management of acquired ataxias focuses on treating the underlying cause.

Non-pharmacological therapeutic options for both acquired and genetic ataxias include symptomatic and multidisciplinary rehabilitation, involving occupational therapy, intensive physiotherapy, and, where available, transcranial magnetic stimulation. Although the effectiveness of these interventions largely depends on the intensity and repetition of functional movements and balance exercises, interactive video game training has shown promise in improving motor abilities even in advanced stages.

Healthcare approaches are both restorative and compensatory. Compensatory aids such as movement decomposition, auditory and visual cues, viscoelastic resistance, computer adaptations (e.g., mouse speed), and walking aids (with or without weights) help maintain or perform activities important to the patient. Restorative approaches focus on repeating specific movements with or without biofeedback, functional movements, and postural control exercises in various environments and situations.

Traditional physical therapy aims to improve postural control and gait and includes physical (re-)conditioning, range-of-motion exercises, muscle strengthening, static and dynamic balance exercises in various positions (e.g., upright kneeling, quadruped, half-kneeling), spinal mobilization, and indoor/outdoor walking. Occupational therapy targets daily living activities such as hygiene, dressing, writing, and eating, and also includes coordination and balance exercises.

Nevertheless, ataxia remains the most treatment-resistant neurological symptom. Given the cerebellum's role in motor learning-particularly error-based learning and adaptation-individuals affected by ataxia often exhibit significant impairments in acquiring both simple and complex motor skills.

Consequently, it is essential to have assessment tools for ataxia that are not only valid and reliable but also sensitive to change. Typically, the evaluation of cerebellar motor syndrome includes five cardinal domains: gait and balance, upper limb coordination, lower limb coordination, speech clarity, and oculomotor control. To understand the differences among currently available scales, a description of the main instruments used to rate the severity of impairment is necessary.

Ataxia Rating Scales

A recent literature review identified 14 instruments and recommended the Friedreich's Ataxia Rating Scale (FARS), the International Cooperative Ataxia Rating Scale (ICARS), and the Scale for the Assessment and Rating of Ataxia (SARA) as the most appropriate tools for evaluating ataxia, excluding condition-specific scales such as the Unified Multiple System Atrophy Rating Scale (UMSARS). However, the four most widely used and studied scales are SARA, ICARS, FARS, and the Brief Ataxia Rating Scale (BARS).

These scales assess signs, symptoms, and the impact of cerebellar ataxia on daily activities, providing a clinical score. Originally developed by clinicians, they have been validated to reflect patients' lived experiences with cerebellar motor syndrome. A recent study confirmed the alignment between spontaneously reported symptoms by patients and caregivers and the concepts measured by these scales.

SARA (Scale for the Assessment and Rating of Ataxia) SARA is the most commonly used scale in both clinical and research settings worldwide. It was preferred over ICARS due to similar clinimetric properties-excellent validity and reliability, with no floor or ceiling effects-but with a shorter administration time. SARA consists of 8 items assessing gait, balance, upper and lower limb coordination, and speech articulation. Each item is scored on an ordinal scale, yielding a total score ranging from 0 (no ataxia) to 40 (severe ataxia).

Developed in 2006 for spinocerebellar ataxia, SARA has since been validated in populations with stroke, Friedreich's ataxia, multiple sclerosis (MS), and lysosomal storage disorders. It demonstrates high reliability: inter-rater (ICC: 0.921-0.98), intra-rater (ICC: 0.952-0.99), and test-retest (ICC: 0.90), with adequate internal consistency (Cronbach's α: 0.89-0.97 depending on population).

Correlations include:

MS: Expanded Disability Status Scale (rho = 0.557) Friedreich's Ataxia: FARS (r = 0.938) All ataxias: Barthel Index (r = -0.63) Stroke: Barthel Index (r = -0.792) In terms of sensitivity to change, for lysosomal storage disorders, an area under the curve (AUC) of 0.82 and a 1-point change is considered clinically significant. For spinocerebellar ataxias, the standardized response mean (SRM) is 0.50, with an average annual score change of 1.38/40 ± 2.8 SD.

A shortened version, the modified-functional SARA (f-SARA), was recently developed by a pharmaceutical group to provide a clinically meaningful measure of disease progression. It appears sensitive enough to detect significant changes over one year, with a 1-point intra-individual threshold . However, SARA remains more precise for tracking disease progression, as item reduction in f-SARA compromises its granularity .

ICARS (International Cooperative Ataxia Rating Scale) Developed in 1997, ICARS includes 19 items across four subcategories: posture and gait disturbances, limb ataxia, dysarthria, and oculomotor disorders. Most items are scored on an ordinal scale, except one binary item assessing saccadic dysmetria. The total score ranges from 0 (no ataxia) to 100 (severe ataxia) .

ICARS has been validated in various populations, including focal lesions, Friedreich's ataxia, chronic alcoholism, and spinocerebellar ataxias. It shows good validity and excellent reliability (inter-rater ICC: 0.95; intra-rater ICC: 0.97), but its 30-minute administration time limits routine use. ICARS is particularly effective in distinguishing mild from moderate ataxia in MS patients (AUC: 0.875) .

BARS (Brief Ataxia Rating Scale) Developed in 2009 as a shortened version of ICARS, BARS includes 5 items focusing on key motor domains: gait, heel-knee test, finger-nose test (scored 0-4), dysarthria, and oculomotor abnormalities. The total score ranges from 0 (no ataxia) to 19 (severe ataxia).

BARS is valid (correlation with SARA: r = 0.91), reliable (inter-rater ICC: 0.91), and sufficiently fast and accurate for clinical use, though it remains underutilized .

FARS (Friedreich's Ataxia Rating Scale)

FARS comprises five subdomains assessing:

(A) Bulbar function (B) Upper limb coordination (C) Lower limb coordination (D) Peripheral nervous system (E) Upright stability Only subdomains B, C, and E are specific to ataxia and overlap with SARA and ICARS. A shortened version of FARS also exists, maintaining excellent clinimetric properties.

Among all these scales, SARA is the most frequently used tool in clinical practice in French-speaking Switzerland, as it has undergone a transcultural validation process and is therefore available in French. However, physiotherapists involved in the rehabilitation of individuals with ataxia encounter limitations when using SARA to assess their patients. Specifically, SARA does not allow for the objectification of fluctuations that therapists observe in clinical settings. Moreover, some patients have reported that SARA scores do not meaningfully reflect their clinical condition .

One possible explanation is that SARA includes global activities such as gait and balance. In this population, improvements in activities are often contingent upon improvements in impairments. The first hypothesis is that it is necessary to improve functions or impairments-according to the terminology of the International Classification of Functioning, Disability and Health (ICF)-in order to impact activity levels. The goal was therefore to develop a scale that evaluates functions, enabling the detection of smaller variations in patients' motor abilities.

A second hypothesis is that more distal and fine motor activities may better capture changes. For example, in a population of individuals with ataxia, the Nine Hole Peg Test (9HPT), which assesses manual dexterity, was found to be more sensitive to change than SARA. Finally, SARA includes only a few global tests for upper and lower limbs, while the trunk is largely absent from the evaluated components. The objective of the new ATLAS scale was thus to address this gap by incorporating trunk assessment, evaluating limbs with greater precision, and including distal motor evaluation.

Another team of clinician-researchers recently sought to go beyond traditional time-based or task-completion measures used in SARA and ICARS, and to include trunk assessment. They developed the Comprehensive Coordination Scale (CCS), which evaluates both performance and movement quality. It consists of six tests assessing motor coordination of the trunk, upper limbs, lower limbs, or their combination: finger-to-nose test, arm-trunk coordination test, finger opposition, interlimb coordination, Lower Extremity Motor Coordination Test (LEMOCOT), and four-limb coordination.

ATLAS, developed by a local team, differs from CCS by including scoring for upper and lower trunk control across different planes, and by evaluating the shoulder, elbow, wrist, hip, knee, and ankle levels distinctly and specifically. Moreover, the final item in CCS-four-limb coordination-is not under cerebellar control and is therefore considered inappropriate for the objectives of our project.

Ataxia Trunk, Lower And upper extremity Scale (ATLAS) The Ataxia Trunk, Lower And upper extremity Scale (ATLAS) was developed by expert physiotherapists in collaboration with the Principle Investigator. The team undertook a process of hierarchical structuring and scoring of clinical tests taught in postgraduate training. These tests are based on the work of Regula Steinlin Egli, a specialist in neurological physiotherapy and author of "Multiple Sklerose verstehen und behandeln".

Steinlin Egli derived these tests from the concept developed by Suzanne Klein-Vogelbach (1909-1996), which advocates for a dynamic and functional analysis of movement (Funktionelle Bewegungslehre - FBL). This concept emphasizes precise observation of functional movements, their segmentation, and active correction through targeted exercises to retrain motor patterns and improve movement efficiency. Special attention is given to posture and the relationship between the trunk and limbs in daily activities.

This functional movement analysis is reflected in the tests presented by Steinlin Egli, an instructor of FBL Klein-Vogelbach, and consequently in the ATLAS scale.

As previously mentioned, scoring was assigned to Steinlin Egli's tests, and variations were created, tested, and validated by expert physiotherapists in ataxia during several quality circle meetings.

The scale is named Ataxia Trunk, Lower, And upper extremity Scale (ATLAS). It includes 20 items: 14 for the trunk, 3 for the lower limbs (LL), and 3 for the upper limbs (UL). Each item is rated on an ordinal scale with 2 to 4 levels. A maximum total score of 64 indicates severe ataxia, while 0 indicates no ataxia. The maximum sub-scores are: trunk - 28, LL - 18, UL - 18, with each side assessed separately.

The content validity of ATLAS was established through observation of ataxic patients, clinical experience of the authors, and discussion and adaptation of the content with specialists in neurological rehabilitation.

The acceptability and feasibility of ATLAS has been tested among patients, members of the quality circle, and the physiotherapy and occupational therapy teams at the Lavigny Institution, as well as the principal investigator.

This scale is an Observer-Administered Clinical Outcomes Assessment (COA) for cerebellar motor syndrome, similar to its counterparts. ATLAS distinguishes itself by focusing on the evaluation of segmental coordination abilities, specifically of the trunk, lower limbs, and upper limbs. It is intended for use primarily by physiotherapists and occupational therapists to monitor their patients over time.

Due to its specific assessment of coordination capacities across different body segments, ATLAS will be particularly useful for physiotherapists. It enables them to set appropriate sub-goals for treatment. For example, if a person with motor symptoms of ataxia wishes to descend stairs independently and safely without using the handrail, the physiotherapist will be able to identify which body segment(s) require targeted intervention in addition to functional training. The scale may indicate, for instance, a deficit in right hip coordination and a need for improved dynamic stabilization of the lower trunk.

Like other scales, ATLAS also allows for reassessment at the end of a specific rehabilitation program or during regular follow-up in the case of hereditary ataxias. While its primary purpose is clinical use, it may also be of interest for research, particularly in studies evaluating the effects of interventions on ataxia.

Project Objectives The main objective of this project is to validate the new ATLAS scale, which assesses cerebellar motor symptoms, with a particular focus on its structural validity. This includes a goal of item reduction. Secondary objectives include evaluating its internal consistency, concurrent validity, and inter-rater reliability.

The target population for this scale includes individuals presenting with cerebellar motor symptoms, whether of hereditary or acquired origin. However, for the purpose of validation, it is necessary to include only individuals whose symptoms are primarily or exclusively cerebellar. Concomitant impairments-such as significant muscle weakness, spasticity, choreic or dystonic movements-could influence test results and compromise the evaluation of each item's validity. Therefore, the aim is to validate the scale in populations with "pure" cerebellar symptomatology, such as those with hereditary ataxia or following a cerebellar or pontine stroke.

ELIGIBILITY:
Inclusion Criteria:

* Be adults
* Be able to provide written informed consent
* Be able to understand and follow simple physical instructions
* Have a diagnosis of genetic or hereditary ataxia, or a cerebellar or pontine stroke (either hemorrhagic or ischemic), confirmed by a neurologist

Exclusion Criteria:

* Muscle group strength < 3 on the Medical Research Council (MRC) scale
* Spasticity > 2 in any muscle on the Modified Ashworth Scale
* Pain > 5 on the Visual Analogue Scale (VAS) in any part of the body

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population of the study consists of individuals with motor impairments of cerebellar origin. These individuals are expected to exhibit typical symptoms of cerebellar dysfunction and, as such, will be found among those with hereditary or genetic ataxia, as well as individuals who have experienced a pontine or cerebellar stroke.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Ataxia Trunk, Lower And upper extremity Scale scores (ATLAS) | Once, at day 1
  The Ataxia Trunk, Lower And upper extremity Scale (ATLAS) includes 20 items: 14 related to the trunk, 3 to the lower limbs (LL), and 3 to the upper limbs (UL). Each item is rated using an ordinal scale ranging from 2 to 4. A maximum total score of 64 indicates severe ataxia, while a score of 0 reflects the absence of ataxia. The maximum subscore for the trunk is 28, for the lower limbs 18, and for the upper limbs 18, with each side assessed separately.

SECONDARY OUTCOMES:
Functional Independence Measure (FIM) | Once, at day 1
  The Functional Independence Measure (FIM) assesses six functional domains using 18 items: Self-care, Sphincter control, Mobility/Transfers, Locomotion, Communication, and Social cognition. These items are grouped into two domains: Motor (13 items) and Cognitive (5 items). Each item is rated on a 7-point Likert scale, where 1 indicates complete dependence requiring total assistance, and 7 indicates complete independence. Assessment can be conducted through interview or direct observation of performance. The total score ranges from 18 to 126 points, with 18 representing complete dependence and 126 representing full independence. Subscores for the Motor and Cognitive domains can also be calculated.
Trunk Impairment Scale 2.0 (TIS 2.0) | Once, at day 1
  Trunk Impairment Scale 2.0 is a shortened form of the Trunk Impairment Scale. The scale consists of 7 tests, each rated using an ordinal scale with 2 or 3 levels (0 to 2), based on observational criteria. It is divided into two categories: Dynamic Sitting Balance (10 points) and Coordination (6 points). Higher scores indicate better functional abilities.
Scale for the Assessment and Rating of Ataxia (SARA) | Once, at day 1
  The Scale for the Assessment and Rating of Ataxia includes 8 items assessing different aspects of ataxia, such as gait, balance, upper and lower limb coordination, and speech articulation. Each item is rated on an ordinal scale, resulting in a total score ranging from 0 (no ataxia) to 40 (severe ataxia).

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Ferchichi-Barbey, Master, Principal Investigator — HESAV School of Health Sciences - Vaud, HES-SO University of Applied Sciences and Arts Western Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Could be shared, platform not yet identified